CLINICAL TRIAL: NCT05087810
Title: Stress and Anxiety Effects on Overactive Bladder
Status: Terminated | Type: Observational
Why Stopped: Change in status - Update June 2024: Upon guidance from the funding source (NIDDK), this record was pdated to an observational study as it was determined not to be an interventional clinical trial.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Elisabeth Sebesta, Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: 211147
Record Dates: First submitted 2021-09-08; First posted 2021-10-21 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Overactive Bladder; Stress, Psychological; Anxiety
MeSH Terms: conditions — Urinary Bladder, Overactive; Stress, Psychological; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects: All subjects will undergo accelerated oral hydration to induce diuresis and then acute psychological stress tasks to induce acute stress. Outcomes will measure changes to perceived bladder sensation in response to acute stress provocation.
  Interventions: Behavioral: Psychological stress induction; Other: Accelerated oral hydration

INTERVENTIONS:
Behavioral: Psychological stress induction — Subjects will undergo acute psychological stress induction by performing mental arithmetic tasks.
Other: Accelerated oral hydration — Participants will drink 2L of fluid in a short period of time to force diuresis and urine production.

SUMMARY:
The purpose of this study is to assess how psychological stress and anxiety relate to bladder sensitivity and to psychological burdens in people with overactive bladder and how this can be measured effectively. UPDATE: June 2024 - Upon guidance from the NIDDK, this record was updated to an observational study as it was determined not to be an interventional clinical trial.

DETAILED DESCRIPTION:
Overactive bladder (OAB) (i.e. urinary urgency, with or without urgency urinary incontinence, frequency, and nocturia) affects 1 in 7 U.S. men and women and results in substantial impairment to quality of life (QOL). To help self-manage and cope with OAB, many people adopt compensatory bladder behaviors, such as restricting fluids, using containment products, strategic planning and mapping restroom access, and even curtailing activities or travel altogether, which further adversely impact QOL. These behaviors may be driven by anxiety and stress related to urinary urgency and incontinence episodes as well as ensuing distress and embarrassment. Prior research has linked anxiety and OAB: up to 40% of women and 30% of men with OAB also have generalized anxiety disorder. The link between stress and OAB is less studied. In animals, experimental stress can cause OAB-like symptoms and behaviors as well as bladder and somatic hypersensitivity. In limited human studies, women with OAB may have greater physiologic and psychologic stress reactivity, and acute stress may exacerbate urinary urgency. However, how stress impacts on the bladder in the context of OAB or what psychological factors drive compensatory behaviors that impair QOL in OAB remain unknown, as there are no highly-controlled studies of anxiety-OAB links. Understanding these relationships would be a critical advance to individualizing care of patients with OAB. The proposed project will comprehensively investigate for the first time how stress, anxiety and OAB interact, including the impacts on bladder sensitivity, urinary symptoms, and compensatory bladder behaviors. The investigators propose a feedforward loop, whereby increased OAB symptoms increase anxiety (via response to coping with stressful situations), which in turn increases OAB symptoms (via increased bladder sensitivity). The study further proposes that compensatory behaviors are driven by anxiety-related learning processes that help perpetuate this relationship. The team will test the hypotheses in a sample of men and women with OAB and healthy controls. Aim 1 will test the hypothesis that acute, experimentally induced psychological stress will be more strongly associated with increased bladder sensitivity in OAB patients than in controls, using a novel bladder sensation meter with oral hydration and stress induction procedures. Aim will test the hypothesis that psychological stress and anxiety will have concurrent and lagged effects on day-to-day urinary symptoms that are stronger in individuals with OAB than in controls, using an ecological momentary assessment approach (7-day electronic diary) to examine prospective associations between everyday perceived stress, anxiety and urinary symptoms. Aim 3 will test the hypothesis that compensatory behaviors (i.e. coping) used at the time of voiding will be associated with subsequent reductions in anxiety levels, using a 3-day sensation-related bladder diary that captures concurrent bladder behaviors and anxiety symptoms as well as lagged symptoms 30 minutes post-void. Delineating these relationships and patterns will allow for identification of potentially modifiable factors or areas for intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, at least 18 years of age
* Cognitive status and English language skills sufficient to complete all study related assessment materials
* Presence of OAB (score of ≥4 on the OAB-V3 awareness tool)
* Urgency predominant urinary incontinence, if incontinence present

Specific entry criteria for control subjects

* Subject to the same inclusion/exclusion criteria, plus:
* Absence of OAB (score of ≤3 on the OAB-V3)
* No urgency-related urinary incontinence

Exclusion Criteria:

* Post void residual urine >150ml
* Need for catheterization, indwelling or intermittent
* Men: uroflow < 10 ml per sec
* Current symptomatic urinary tract infection that has not resolved
* Comorbid neurological conditions, including spinal cord injury, systemic neurologic illnesses (i.e. multiple sclerosis, Parkinson's disease) or central nervous system disease (i.e. brain tumor, stroke) thought to impact bladder function
* Iatrogenic (i.e. post-surgical) or non-iatrogenic obstructive conditions (i.e. pelvic organ prolapse greater than stage 2, urethral stricture, benign prostatic enlargement)
* Prior pelvic irradiation
* Current or prior bladder malignancy
* Confirmed diagnosis of Interstitial Cystitis
* Hematuria without a clinically appropriate evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This prospective observational cohort study will recruit individuals with overactive bladder and age/sex matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Bladder stress reactivity | 30 minutes
  Changes to bladder sensation prompted by acute psychological stress tasks as measured by degree of perception of bladder fullness (100 point scale)

SECONDARY OUTCOMES:
Systolic blood pressure responses | 30 minutes
  Changes to non-invasive systolic blood pressure prompted by psychological stress tasks.
Diastolic blood pressure response | 30 minutes
  Changes to non-invasive diastolic blood pressure prompted by psychological stress tasks.
Heart rate response | 30 minutes
  Changes to non-invasive heart rate prompted by psychological stress tasks.

CONTACTS AND LOCATIONS:
Overall Officials: William S Reynolds, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No